CLINICAL TRIAL: NCT04048655
Title: Reversal of Neuromuscular Blockade During the General Anaesthesia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R19095M
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Neuromuscular Blockade
Keywords: neuromuscular blockade; neostigmine; muscle relaxation; train of four; rocuronium
MeSH Terms: interventions — Neostigmine

STUDY DESIGN:
Intervention Model Description: Single group with same study protocol to asses the incidence of postrecovery relaxation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Other): Single arm and everyone gets the same treatment according the protocol
  Interventions: Drug: Neostigmine, Combinations

INTERVENTIONS:
Drug: Neostigmine, Combinations — All patients have neostigmine induced recovery of neuromuscular block.

SUMMARY:
There are individual reports indicating that after the reversal of nondepolarizing neuromuscular blockade with neostigmine, some patients starts to relax spontaneously again after the tof ratio has already recovered to the safe level (>90%).

The mechanism behind this in not well understood, and the incidence of the phenomenon is unclear. In this study the investigators try to determine the incidence of the aforementioned postrecovery relaxation.

DETAILED DESCRIPTION:
There are individual reports indicating that after the reversal of nondepolarizing neuromuscular blockade with neostigmine, some patients start to relax spontaneously again after the tof ratio has already recovered to the safe level (90%). The mechanism behind this in not well understood and the incidence of the phenomenon is unclear.

The aim of this study is to monitor the reversal of rocuronium induced neuromuscular blockade with neostigmine. The neuromuscular blockade is monitored with train of four stimulations using electromyography. After the reversal agent is given and train of four ratio has recovered to the level of 90%, the neuromuscular blockade is monitored another 30min to see if tof ratio starts to spontaneously fall again under the 90%. If aforementioned postrecovery relaxation happens, the investigators are able to calculate the incidence of the phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery requiring general anaesthesia
* Surgery is assumed to last more than 45 minutes
* Body mass index less than 35kg/ m²

Exclusion Criteria:

* Disease of central nervous system
* Trauma of central nervous system
* Disease affecting peripheral nervous system
* Medication affecting peripheral nervous system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postrecovery relaxation | 30 minutes
  Number of patients (if any) with postrecovery relaxation divided by a number of all patients

CONTACTS AND LOCATIONS:
Overall Officials: Maija Kalliomäki, Docent, Study Director — Tampere University Hospital; Jarno Salminen, Licenciate, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland